CLINICAL TRIAL: NCT07015580
Title: The Characteristics of Oral Microbiota in Chronic Pancreatitis and Autoimmune Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, ZOU DUOWU, Director of Gastroenterology Department, Ruijin Hospital
Other Study IDs: RuijinH202538
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Oral Microbiota; Pancreatitis; Pancreatic Cancer
MeSH Terms: conditions — Pancreatitis; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- chronic pancreatitis: Clinical data including medical history, clinical symptoms, imaging examination, laboratory examination will be collected. 3-5ml saliva sample of every patients will be collected for 16S rRNA sequencing of oral microbiota.
  Interventions: Other: 16S rRNA sequencing
- autoimmune pancreatitis: Clinical data including medical history, clinical symptoms, imaging examination, laboratory examination will be collected. 3-5ml saliva sample of every patients will be collected for 16S rRNA sequencing of oral microbiota.
  Interventions: Other: 16S rRNA sequencing
- pancreatic cancer: Gender, age (± 5 years), smoking and drinking are matched with patients with chronic pancreatitis. Clinical data including medical history, clinical symptoms, imaging examination, laboratory examination will be collected. 3-5ml saliva sample of every patients will be collected for 16S rRNA sequencing of oral microbiota. considering sugery or endoscopy may change the oral microbiota, the saliva sample will be collected in pantients with suspected pancreatic cancer. Only pantients with pathologically confirmed pancreatic cancer will be inclueded in final analysis
  Interventions: Other: 16S rRNA sequencing
- healthy control: Gender, age (± 5 years), smoking and drinking are matched with patients with chronic pancreatitis. 3-5ml saliva sample of every participant will be collected for 16S rRNA sequencing of oral microbiota.
  Interventions: Other: 16S rRNA sequencing

INTERVENTIONS:
Other: 16S rRNA sequencing — Clinical data including medical history, clinical symptoms, imaging examination, laboratory examination will be collected. 3-5ml saliva sample of every patients will be collected for 16S rRNA sequencing of oral microbiota.

SUMMARY:
There are more than 700 different bacteria colonized in human oral cavity, which are collectively referred to as oral microbiota. Emerging evidence suggests that oral microbiota plays a series of important roles in human health, such as immune response, carcinogen metabolism and nutrient digestion. The changes of oral microbiota composition are closely related to the occurrence and development of pancreatic diseases. Previous studies have found that there are dense bacterial biofilms in the pancreatic duct of patients with calcified pancreatitis, including oral bacterial types. However, most studies only focused on the changes of gut microbiota in patients with chronic pancreatitis, and there were lack of research and description on the changes of oral microbiota in patients with chronic pancreatitis. In this study, we will extract and sequence bacterie's full-length 16S rRNA to describe the characteristics of oral microbiota in patients with chronic pancreatitis, confirming that there are changes in oral microbiota in patients with chronic pancreatitis, and compare the differences of oral microbiota in patients with chronic pancreatitis, pancreatic cancer and autoimmune pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* A dated and signed informed consent form cooperate to complete sample collection

Exclusion Criteria:

* Previous digestive system surgery; During pregnancy or lactation; Complicated with infectious diseases, malignant tumors or other digestive system diseases (such as inflammatory bowel disease, irritable bowel syndrome, abdominal diseases, gastroesophageal reflux, etc.); Antibiotics and immunosuppressive drugs were used within 30 days before sampling; Those who take probiotics daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic pancreatitis or autoimmune pancreatitis or pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
characteristic of oral microbiota in patients with chronic pancreatitis | From enrollment to the end at 2 weeks
  Species composition of oral microbiota in pantients chronic pancreatitis

SECONDARY OUTCOMES:
Differences in oral microbiota profiles between chronic pancreatitis and autoimmune pancreatitis, pancreatic cancer healthy controll. | From enrollment to the end at 2 weeks
  compare the alpha diversity and beta diversity of different groups. Alpha diversity is an index used to reflect the richness and evenness within a sample.Beta diversity is an indicator of species richness and evenness among samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterolog, Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai, China, China